CLINICAL TRIAL: NCT02825680
Title: Learn, Engage, Act, Process (LEAP) for Personalized Weight Management Support (QUE 15-286)
Brief Title: Learn, Engage, Act, Process (LEAP) for MOVE!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 16-004
Record Dates: First submitted 2016-05-12; First posted 2016-07-07 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: Weight Loss; Body Weight Maintenance; Quality Improvement
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced NCP Support (Active Comparator): Teams at facilities who expressed interest in being in the trial but who are not randomly assigned to the experimental arm will be in the active comparator arm. These facilities will receive enhanced support from NCP.
  Interventions: Other: Enhanced NCP Support
- LEAP Intervention (Experimental): Cohorts of 6 facilities, who expressed interest in being in the trial, will be randomly selected each quarter, as guided by the stepped-wedge trial design protocol, to participate in LEAP. These facilities will also receive the same enhanced NCP support as received by the active comparator arm.
  Interventions: Other: Enhanced NCP Support; Other: LEAP

INTERVENTIONS:
Other: Enhanced NCP Support — NCP is a central policy office that provides support to MOVE! program teams through monthly phone calls and technical assistance. Facilities will also have access to the audit and feedback process and barrier buster tool
Other: LEAP — The Learn. Engage. Act. Process (LEAP) intervention relies on virtual (phone and online) coaching based on the IHI Model for Improvement, an online learning platform for clinician teams to share ideas and progress, an audit and feedback process, and a barrier buster tool.
  Arms: LEAP Intervention

SUMMARY:
The overall goal of this project is to test whether the Learn. Engage. Act. Process (LEAP) intervention helps teams within the Veterans Health Administration's (VHA) local MOVE! group weight management programs be more in line with guidance. Forty-eight sites will be randomized to the LEAP intervention, which is a virtually delivered program that relies on the Institute for Healthcare Improvement (IHI) Model for Improvement, an online learning platform for clinician teams to share ideas and progress, an audit and feedback process, and a barrier buster tool. The LEAP intervention will be compared to active support that is provided to all VA MOVE! programs by the National Center for Health Promotion and Disease Prevention (NCP). The investigators will compare whether participation in LEAP results in engaging more Veterans in the MOVE! weight management program compared to facilities not participating in LEAP. The investigators will also collect information to understand what components of LEAP worked best and how to scale up so more teams can participate in LEAP.

DETAILED DESCRIPTION:
The Veterans Affairs (VA) National Center for Health Promotion and Disease Prevention (NCP) first disseminated MOVE! weight management program guidance in 2006. Program guidance was updated in 2014, which is expected to increase engagement and improve outcomes. However, variation in local programs is high. The overall goal of this project is to test the Learn. Engage. Act. Process (LEAP) intervention to work with teams virtually, to build skills in implementing program improvements. Forty-eight sites will be randomized to the LEAP intervention using a stepped-wedge trial design. LEAP is a virtually delivered program that relies on the IHI Model for Improvement, an online learning platform for clinician teams to share ideas and progress, an audit and feedback process, and a barrier buster tool. The LEAP intervention will be compared to active support provided by NCP to all local VA MOVE! teams. The investigators will compare whether teams participating in LEAP have MOVE! programs that engage more Veterans compared to facilities not participating in LEAP. The investigators will also collect information to understand which components of LEAP worked best and how to scale up and implement LEAP more broadly. The project aims are:

Aim 1: To develop three core products to enhance NCP support to Veterans Affairs Medical Centers (VAMCs) and to pilot LEAP in three VAMCs.

H1: Dissemination of products to enhance NCP support will improve MOVE! outcomes.

Aim 2: To determine effectiveness of LEAP plus enhanced NCP support (LEAP+NCP) versus enhanced NCP support alone.

H2: VAMCs with LEAP+NCP will have better MOVE! group outcomes than VAMCs with enhanced NCP support alone.

Aim 3: To conduct formative and cost evaluations to refine design of LEAP and inform future scaling-up of LEAP.

ELIGIBILITY:
Inclusion Criteria:

* Unit of randomization is facility.
* MOVE! group program in a VA Medical Center.
* MOVE! coordinators at medical centers who express interest in participating in the trial prior to the first cohort randomization.

Exclusion Criteria:

* Unit of randomization is facility.
* Facilities that are not a medical center e.g., community-based outpatient clinic, Veteran service center

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura J. Damschroder, MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Primary outcome is based on data aggregated to the facility level. Thus, this question is N/A.

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced NCP Support: Teams at facilities who expressed interest in being in the trial but who are not randomly assigned to the experimental arm will be in the active comparator arm. These facilities will receive enhanced support from the National Center for Health Promotion and Disease Prevention (NCP).
  Enhanced NCP Support: NCP is a central policy office that provides support to MOVE! program teams through monthly phone calls and technical assistance. Facilities will also have access to the audit and feedback process and barrier buster tool
- LEAP Intervention: Cohorts of 6 facilities, who expressed interest in being in the trial, will be randomly selected each quarter, as guided by the stepped-wedge trial design protocol, to participate in LEAP. These facilities will also receive the same enhanced NCP support as received by the active comparator arm.
  Enhanced NCP Support: NCP is a central policy office that provides support to MOVE! program teams through monthly phone calls and technical assistance. Facilities will also have access to the audit and feedback process and barrier buster tool
  LEAP: The Learn. Engage. Act. Process (LEAP) intervention relies on virtual (phone and online) coaching based on the Institute for Healthcare Improvement (IHI) Model for Improvement, an online learning platform for clinician teams to share ideas and progress, an audit and feedback process, and a barrier buster tool.
Period: Overall Study
Arm/Group | Enhanced NCP Support | LEAP Intervention
Started | 82 | 55
Completed | 82 | 39
Not Completed | 0 | 16

BASELINE CHARACTERISTICS:
Population: This study did not collect data about individual patients. The unit of randomization for this study was VA Medical Centers. The unit of measurement is facility aggregated data.
Groups:
- Enhanced NCP Support: Teams at facilities who expressed interest in being in the trial but who are not randomly assigned to the experimental arm will be in the active comparator arm. These facilities will receive enhanced support from the National Center for Health Promotion and Disease Prevention (NCP).
  Enhanced NCP Support: NCP is a central policy office that provides support to MOVE! program teams through monthly phone calls, online tools and resources, and technical assistance. Facilities will also have access to a customized "cube" of administrative data including sessions delivered, weight outcomes, and levels of participation for all Veterans Health Administration (VHA) MOVE! programs.
- LEAP Intervention: Cohorts of 6 facilities, who expressed interest in being in the trial, will be randomly selected each quarter, as guided by the stepped-wedge trial design protocol, to participate in LEAP. These facilities will also receive the same enhanced NCP support as received by the active comparator arm.
  Enhanced NCP Support: NCP is a central policy office that provides support to MOVE! program teams through monthly phone calls, online tools and resources, and technical assistance. Facilities will also have access to a customized "cube" of administrative data including sessions delivered, weight outcomes, and levels of participation for all VHA MOVE! programs.
  LEAP: The Learn. Engage. Act. Process (LEAP) intervention relies on virtual (phone and online) coaching based on the Institute for Healthcare Improvement (IHI) Model for Improvement, an online learning platform for clinician teams to share ideas and progress, an audit and feedback process, and a barrier buster tool.
- Total: Total of all reporting groups
Arm/Group | Enhanced NCP Support | LEAP Intervention | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Rate of MOVE! Visits Per 1000 Candidate Veterans
Description: Rate is calculated as aggregate number of MOVE! group visits per facility divided by aggregate count of candidate Veterans living w/in 40 miles multiplied by 1000. This will include facility level aggregated number of MOVE! group visits at rolling prospective 6 month time periods after the end of each stepped-wedge cohort timeframe. Time periods are rolling based on stepped-wedge trial design. Data will be extracted from the Corporate Data Warehouse (CDW).
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Rate of MOVE! Visits per 1000 Candidate
Groups:
- LEAP Intervention: Cohorts of 6 facilities, who expressed interest in being in the trial, will be randomly selected each quarter, as guided by the stepped-wedge trial design protocol, to participate in LEAP. These facilities will also receive the same enhanced NCP support as received by the active comparator arm.
  Enhanced NCP Support: NCP is a central policy office that provides support to MOVE! program teams through monthly phone calls and technical assistance. Facilities will also have access to the audit and feedback process and barrier buster tool
  LEAP: The Learn. Engage. Act. Process (LEAP) intervention relies on virtual (phone and online) coaching based on the IHI Model of Change, an online learning platform for clinician teams to share ideas and progress, an audit and feedback process, and a barrier buster tool
Arm/Group | Enhanced NCP Support | LEAP Intervention
Number analyzed (Participants) | 82 | 55
Rate of MOVE! Visits per 1000 Candidate
  Before LEAP | 4.504 [4.267 to 4.742] | 4.853 [4.555 to 5.150]
  After LEAP | 4.824 [4.414 to 5.233] | 5.061 [4.677 to 5.445]
Statistical Analysis 1: Comparison: Enhanced NCP Support vs LEAP Intervention; This analysis compares reach within the pre-intervention timeframe versus the post-intervention timeframe for each LEAP (intervention) and control case. Intention to treat analysis was used; all participating facilities randomized to the LEAP (intervention) arm were included whether or not they completed the intervention; Test type: Superiority; p = .011, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: This study did not collect data about individual patients. The unit of randomization for this study was VA Medical Centers. Participants in this study were a team of healthcare providers from the group MOVE! weight management program at each participating VA Medical Center.
Description: Participants for this study were VA facilities and not individual patients.
Arm/Group | Enhanced NCP Support | LEAP Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a pragmatic trial. Our main outcome measure relied on administratively collected data. Additionally, the causal pathway that leads from LEAP coaching to reach outcomes is likely impacted by unmeasured influences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02825680/Prot_SAP_000.pdf